CLINICAL TRIAL: NCT02083341
Title: Effects of External Vibration on Voice Quality in Muscle Tension Dysphonia Patients and Classically Trained Singers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VVT-01; AHSC AFP Innovation Fund (Other Grant/Funding Number: MOHLTC Ontario)
Record Dates: First submitted 2014-03-05; First posted 2014-03-11 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Dysphonia; Singing
MeSH Terms: conditions — Dysphonia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Muscle tension dysphonia - treatment (Experimental): external vibration device. A prospective, randomized, placebo controlled, single blinded study design will be used to investigate the effects of an external vibration device on voice acoustic parameters and perceptual in MTD patients and singers. The external vibration device to be investigated is the Lelo® Siri vibrator. The external vibration therapy sessions, and pre and post acoustic recordings will be conducted by a SLP.
  Interventions: Device: Lelo® Siri vibrator
- Muscle tension dysphonia - Sham (Sham Comparator): external vibration device - sham. A prospective, randomized, placebo controlled, single blinded study design will be used to investigate the effects of an external vibration device on voice acoustic parameters and perceptual in MTD patients and singers. The external vibration device to be investigated is the Lelo® Siri vibrator. The external vibration therapy sessions, and pre and post acoustic recordings will be conducted by a SLP. Lelo® Siri vibrator with vibration component removed.
  Interventions: Device: Lelo® Siri vibrator with vibration component removed
- Classically trained singers (Experimental): external vibration device. A prospective, randomized, placebo controlled, single blinded study design will be used to investigate the effects of an external vibration device on voice acoustic parameters and perceptual in MTD patients and singers. The external vibration device to be investigated is the Lelo® Siri vibrator. The external vibration therapy sessions, and pre and post acoustic recordings will be conducted by a SLP.
  Interventions: Device: Lelo® Siri vibrator
- Classically trained singers - Sham (Sham Comparator): external vibration device - sham. A prospective, randomized, placebo controlled, single blinded study design will be used to investigate the effects of an external vibration device on voice acoustic parameters and perceptual in MTD patients and singers. The external vibration device to be investigated is the Lelo® Siri vibrator. The external vibration therapy sessions, and pre and post acoustic recordings will be conducted by a SLP. Lelo® Siri vibrator with vibration component removed.
  Interventions: Device: Lelo® Siri vibrator with vibration component removed

INTERVENTIONS:
Device: Lelo® Siri vibrator — external vibration device
  Arms: Classically trained singers; Muscle tension dysphonia - treatment
Device: Lelo® Siri vibrator with vibration component removed — external vibration device - sham
  Arms: Classically trained singers - Sham; Muscle tension dysphonia - Sham

SUMMARY:
Muscle tension dysphonia (MTD) is a disabling voice disorder which causes severe voice change, neck pain, and voice fatigue. Current therapy modalities to treat these disorders include multiple visits to a qualified speech language pathologist (SLP) for rehabilitation with voice exercises and focused laryngeal/neck massage. Access to these services is difficult with long waitlists and often not covered by current public health insurance or locally available to many patients in Ontario. The goal of this study is to demonstrate a reduction in symptoms and improvement in vocal function by applying an external vibration device to key sites (e.g. jaw, neck, skull base) commonly identified as a source of abnormal muscle tension and injury in certain voice disorders, specifically MTD.

This study will also investigate the effect of external vibration on the voice quality in classically trained singers (CTSs). Certain desirable acoustic qualities in a singers' voice are only accessible when the larynx and its extrinsic muscles are in a relaxed state. Muscle misuse and vocal strain are common problems in performers, which can result in conditions that require surgery and speech therapy, and may lead to a loss of income. Similar to vocal warm up exercises which contribute to the prevention of vocal injury, external vibration is expected to improve muscle perfusion in an acute setting and may have a direct effect on vocal fold cover viscosity.

Both study groups will be randomized to receive either the external vibration device or a sham device. The sham device looks identical to the experimental device but has the vibration component removed.

DETAILED DESCRIPTION:
Muscle tension dysphonia is primarily treated with voice therapy with a qualified SLP. One of the key therapy tools for MTD is laryngeal extrinsic muscle massage along with voice and respiratory exercises. Access to these specialized services is difficult due to limited expertise and travel distance. The goal of this study is to demonstrate a reduction in symptoms and improvement in vocal function by applying an external vibration device to key sites (e.g. jaw, neck, skull base) commonly identified as a source of abnormal muscle tension and injury in certain voice disorders, specifically MTD. If the study shows a demonstrable benefit, patients would be trained to self administer the treatment along with a home program of therapy exercises. This novel therapy would improve delivery of care and allow speech therapy services to be more widely accessible with reduced number of therapy sessions required. The potential long term effects would be to decrease wait times to access these specialized services and lessen the need for return visits due to symptom recurrence.

The second part of this study is to investigate the effect of external vibration on the voice quality in CTSs. Certain desirable acoustic qualities in a singers' voice are only accessible when the larynx and its extrinsic muscles are in a relaxed state. Muscle misuse and vocal strain are common problems in performers, which can result in conditions that require surgery and speech therapy, and may lead to a loss of income. Similar to vocal warm up exercises which contribute to the prevention of vocal injury, external vibration is expected to improve muscle perfusion in an acute setting and may have a direct effect on vocal fold cover viscosity.

ELIGIBILITY:
MTD Inclusion Criteria:

* Diagnosed with primary MTD

MTD Exclusion Criteria:

* Active smoker
* Currently receiving voice therapy from a SLP
* Currently receiving botox injections
* Past laryngeal surgery

CTS Inclusion Criteria:

* Professional or semi-professional classical singer
* Third year university performance major or greater CTS Exclusion Criteria
* Active smoker
* Known voice disorders
* Past laryngeal surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-08; Primary Completion 2016-01-15 (Actual); Study Completion 2016-01-15 (Actual)

PRIMARY OUTCOMES:
jitter | measured at beginning and end of 1 hour study visit (before and after external vibration therapy)
  acoustic measurement from voice recordings

SECONDARY OUTCOMES:
shimmer | measured at beginning and end of 1 hour study visit (before and after external vibration therapy)
  acoustic measurement from voice recordings
signal to noise ratio | measured at beginning and end of 1 hour study visit (before and after external vibration therapy)
  acoustic measurement from voice recordings
fundamental frequency | measured at beginning and end of 1 hour study visit (before and after external vibration therapy)
  acoustic measurement from voice recordings
singing power ratio (singer group only) | measured at beginning and end of 1 hour study visit (before and after external vibration therapy)
  acoustic measurement from voice recordings; captured for the singer group only

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Anderson, MD, FRCS(C), Principal Investigator — Chief, Department of Otolaryngology - Head and Neck Surgery
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Anderson J, DeLuca M, Haines ME, Merrick G. Immediate Effects of External Vibration vs Placebo on Vocal Function Therapy in Singers: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2018 Mar 1;144(3):187-193. doi: 10.1001/jamaoto.2017.2679. PMID 29270622